CLINICAL TRIAL: NCT04938063
Title: Association Between Functional Impairment and Parenting Stress Among Children Diagnosed with Diplegic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed fekry ibrahim salman, Principal Investigator, Cairo University
Other Study IDs: Fekry_phd
Record Dates: First submitted 2021-06-18; First posted 2021-06-24 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy; Parent-Child Relations
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cerebral palsy children: Sample size estimation was carried out to determine the recruited number of the diplegic CP children from the outpatient clinic at the Faculty of Physical Therapy, Cairo University, Physical Therapy Department at the National Institute of Neuromotor Disorder, Abu El-Reesh Hospital, and private physiotherapy clinics. The age of patients will range from 18 months to 5 years old. Both sexes will participate in this study
  Interventions: Other: Assessing the correlation between Functional Impairment and Parenting Stress

INTERVENTIONS:
Other: Assessing the correlation between Functional Impairment and Parenting Stress — Association Between Functional Impairment and Parenting Stress Among Children Diagnosed With Diplegic Cerebral Palsy

SUMMARY:
1. To find out the relation between the severity of ADL limitation in diplegic CP children and the level of parents' stress.
2. To detect the correlation between the PS level to the different domains of ADL limitation.
3. To determine the substantial factors that underlying the parents' stress of those diplegic CP children.

DETAILED DESCRIPTION:
The health and well-being of children are intimately related to their parents' physical, emotional and social health in addition to child-rearing practices. The way parents of CP children deal with their stress may adversely affect their parenting ability, which in turn leads to difficulties for the child, which may lead to more parenting stress. The extent to which parents of CP children adjust and the resources to meet the needs of their children is of primary concern to professionals working in children's healthcare.

To support parents, it is important to determine the level of independence of diplegic CP children in their daily lives. This is necessary to identify predictors of their stress, which may be a mentally debilitating factor in their lives. In return, it may support us as physiotherapists to make more informed decisions about treatment planning, as well as facilitate conversations with parents around identifying sources of stress and developing healthy coping strategies that lead to a better quality of life for their children. Finally, this will have a direct positive impact on the children's abilities

ELIGIBILITY:
Inclusion Criteria:

* Diplegic CP children.
* Their age ranges from 18 months to five years old.
* All levels of GMFCS will be included.
* Both sexes will be included.
* All children were medically and clinically stable.
* Parents must be able to write and read.

Exclusion Criteria:

* Diplegic CP children, who might have one or more of the following:

  * History of chronic cardiac or chest disease.
  * Any behavioral disorders.
  * Current hospitalization for urgent medical reasons.
  * Significant visual or auditory impairment.
  * Previous history of Botox injection within last six months.

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sample size estimation was carried out to determine the recruited number of the diplegic CP children from the outpatient clinic at the Faculty of Physical Therapy, Cairo University, Physical Therapy Department at the National Institute of Neuromotor Disorder, Abu El-Reesh Hospital, and private physiotherapy clinics. The age of patients will range from 18 months to 5 years old. Both sexes will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Assessing the change in parent stress | Baseline only
  It will be assessed by using the approved Arabic version of the Parent stress index. The parent will be asked to read each statement carefully and focus on each statement and circle the one that best suites his psychological state concerning his child. Parents should respond by circling SA (strongly agree), A (agree), NS (not sure), D (disagree), SD (strongly disagree). They should circle only one response per item, and make an "X" through the response if it needs to be changed. Parents must not erase any answers. Parent must be Encouraged to answer all the items.
Assessing the change in children's quality of life | Baseline only
  It will be assessed by The Pediatric Quality of Life Inventory™ (PedsQL™) Family Impact Module version 2 It is composed of parent proxy-report forms obtainable in numerous international languages including Arabic. The Arabic version of the PedsQL™ Family Impact Module version 2.0 is a parent report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family .It consists of 36 items comprising 8 dimensions. It includes 6 subscales measuring parents' self-reported functioning: Physical Functioning (6 items), Emotional Functioning (5items), Social Functioning (4 items), Cognitive Functioning (5 items), Communication (3 items) and Worry (5 items); as well as 2 subscales measuring parent- reported family functioning: Daily Activities (3 items) and Family Relationships (5 items)
Assessing the change in children's activities of daily living | Baseline only
  It will be carried out by using self-care domain (eating, grooming, bathing, dressing upper and lower body and toileting), transfer and locomotion domains of the WeeFIM. Assessment should be performed by direct observing the child. However, when direct observation is not possible, interviewing parents who are familiar with the child's everyday activities is crucial

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Fekry, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic - Faculty of Physical Therapy - Cairo University, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No